CLINICAL TRIAL: NCT06461143
Title: Evaluation of the Efficacy of Computerized Intraosseous Local Anesthesia System in Children With Molar Incisor Hypomineralization
Brief Title: Intraosseous Local Anesthesia System in Children With Molar Incisor Hypomineralization
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The dentist who was taking care of the study's patients stopped working for a while because she went on maternity leave.
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Yelda Kasımoğlu, Assoc. Prof., Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-AKD-97
Record Dates: First submitted 2024-06-04; First posted 2024-06-14 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Molar Incisor Hypomineralization; Hypersensitivity; Composite Restoration
Keywords: dental pain; dental anxiety
MeSH Terms: conditions — Molar Hypomineralization; Hypersensitivity; Toothache

STUDY DESIGN:
Intervention Model Description: Group 1: Intraosseous anesthesia (n=40) Group 2: lnferior alveolar nerve block (n=40)
  Individuals suitable for split-mouth design will be assigned to the opposite anesthesia arm, and their second teeth will be treated and measured.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intraosseous anesthesia (Experimental): Computerized intraosseous anesthesia will be applied to the mandibular first molars of 40 patients.
  Interventions: Drug: %4 articaine with 1:200 000 adrenaline
- Inferior alveolar nerve block (Active Comparator): Conventional inferior alveolar block anesthesia will be applied to the mandibular first molars of 40 patients.
  Interventions: Drug: %4 articaine with 1:200 000 adrenaline

INTERVENTIONS:
Drug: %4 articaine with 1:200 000 adrenaline — For intraosseous anesthesia SleeperOne5 device is going to be used.

SUMMARY:
The goal of this clinical trial is to compare in effectiveness of intraosseous anesthesia and inferior alveolar block anesthesia in children with molar incisor hypomineralization (MIH). The main question it aims to answer are:

- Is intraosseous anesthesia is more effective in pain control when restoring teeth with MIH?

DETAILED DESCRIPTION:
The anxiety experienced by pediatric patients is one of the biggest problems that dentists encounter in practice and is closely related to their current oral health. Studies have shown that dental anxiety depends on many factors, but the pain that is thought to occur during the procedure is one of the most important reasons for the formation of dental anxiety. Painful dental procedures cause anxiety, and anxiety prolongs the duration and increases the severity of the pain felt. For this reason, coping with dentist anxiety at an early age and practices that will enable painless dental treatment in pediatric patients should be emphasized. Behavioral guidance techniques and pain management are used to minimize the pain felt during dental treatment.

Various strategies, devices or techniques have been developed to reduce or eliminate pain occurring during local anesthesia injection. Intraosseous injection is an anesthesia with a high success rate. Anesthesia begins in a short time following the injection, it does not cause numbness in the tongue-lips-cheek, there is almost no injection pain, and less anesthetic solution is used compared to traditional nerve block techniques.

Situations that cause dental anxiety in pediatric patients include children with hypersensitive teeth. Molar incisor hypomineralization (MIH) is a qualitative developmental enamel defect affecting at least one permanent molar. The color of these defects can vary from white to yellow and brown, and especially in severe cases, enamel destruction may occur after application. MIH; dental hypersensitivity is among the most complicated cases that require management of various clinical difficulties in pediatric dentistry, such as failure to provide adequate analgesia/anesthesia, increased risk of carious lesion formation, increased dental anxiety, and increased aesthetic anxiety.

MIH continues to be a subject that continues to be researched in pediatric dentistry. Pediatric dentists encounter difficulties in providing adequate depth of anesthesia in restorative treatments, especially in MIH accompanied by hypersensitivity. This thesis study aims to examine the effect of intraosseous anesthesia on procedural pain in patients with MIH.

As a result of the literature review, the following hypothesis was put forward: There is no significant difference in terms of pain perception between intraosseous anesthesia and traditional metal syringe anesthesia in children with MIH.

ELIGIBILITY:
Inclusion Criteria:

* Individuals applying the Department of Pedodontics, Istanbul University Faculty of Dentistry,
* Systemically healthy,
* Without any allergies,
* Having at least one mandibular first molar with molar incisor hypomineralization (MIH),
* Treatment need index 2 and 4,
* Having a radiographically advanced decay lesion involving dentin (outer ½),
* Possessing sufficient cooperation skills (Frankl scale 3 and 4),
* Between the ages of 6-8,
* Both male and female volunteers will be included.

Exclusion Criteria:

-

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2024-08-21 (Actual); Primary Completion 2026-04-24 (Estimated); Study Completion 2026-05-24 (Estimated)

PRIMARY OUTCOMES:
Wong-Baker FACES Pain Rating Scale | To be measured 2 times on the day of treatment: 1. After local anesthesia application 2. After restoration
  Patient-reported pain. The scale contains a series of six faces ranging from a happy face at 0 to indicate "no hurt" to a crying face at 10 to indicate "hurts worst."

SECONDARY OUTCOMES:
Frankl behaviour rating scale | To be measured 3 times on the day of treatment: 1. Before local anesthesia 2. During local anesthesia 3. During whole treatment
  Behaviour assessment. The Frankl scale is an ordinal scale with 4 ratings used to describe a child's behavior from definitely negative (1), negative (2), positive (3), and definitely positive (4).
Pulse rate | To be measured 3 times on the day of treatment: 1. Before local anesthesia 2. After local anesthesia 3. After restoration
  Pulse rate
Blood pressure | To be measured 3 times on the day of treatment: 1. Before local anesthesia 2. After local anesthesia 3. After restoration
  Blood pressure
MCDAS(f) Turkish version | To be measured 2 times on the day of treatment: 1. In the waiting room before treatment 2. After treatment
  Dental anxiety. Scores on the MCDAS(f) scale may range from 8 to 40, with scores below 19 indicating absence of state anxiety, scores higher than 19 indicating the pres- ence of state anxiety and scores higher than 31, in- dicating severe phobic disorder.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Faculty of Dentistry, Department of Pedodontics, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Can be shared upon the request.